CLINICAL TRIAL: NCT06226454
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Single- and Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Oral VX-993 in Healthy Adult Subjects
Brief Title: A Phase 1 Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics, of VX-993
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX23-993-003
Record Dates: First submitted 2023-12-20; First posted 2024-01-26 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Single Ascending Dose (SAD) (Experimental): Participants will be randomized to receive a single dose of different dose levels of VX-993.
  Interventions: Drug: VX-993
- Part A: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-993.
  Interventions: Drug: Placebo
- Part B: Multiple Ascending Dose (MAD) (Experimental): Participants will be randomized to receive multiple doses of different dose levels of VX-993. The dose levels will be determined based on the data from Part A.
  Interventions: Drug: VX-993
- Part B: Placebo (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-993.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VX-993 — Suspension for oral administration.
  Arms: Part A: Single Ascending Dose (SAD); Part B: Multiple Ascending Dose (MAD)
Drug: Placebo — Suspension for oral administration.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of VX-993 at different doses in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Nonsmoker or ex-smoker for at least 3 months before the first study drug dose

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption, distribution, metabolism, or excretion

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 16
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 43

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-993 | Day 1 up to Day 16
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-993 | Day 1 up to Day 16
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-993 | Day 1 up to Day 43
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-993 | Day 1 up to Day 43
Part B: Pain Tolerance Threshold (PTT) for the Cold Pressor Test | Day 1 up to Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing